CLINICAL TRIAL: NCT06059599
Title: Active Informed Consent: a New Solution to Improve and Objectively Test the Patient Understanding of Complex Surgical Procedures Proposals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CIA21
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Spine Disease; Urologic Diseases
MeSH Terms: conditions — Spinal Diseases; Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active informed consent (Experimental): The experimental group will be prepared for the surgery through the new information tools, a video will be administered with information about the various surgical possibilities, graphics and animations in order to direct the patient toward a more informed choice. Next, an interview with the surgeon will be arranged for the patient and care givers to be listened to and guided through the use of 3D-printed models into the best decision for the individual case (Shared Decision Making - SDM). Having decided on the surgery, patients with similar surgical programs will be guided in educational programs to reinforce information, understanding and long-term retention of the concepts learned. The course will conclude with a second interview with the surgeon and the signing of the standard informed consent.
  Interventions: Other: active informed consent
- Traditional informed consent (No Intervention): The control group of patients will be informed about the surgery according to standard practices. As per standard practice, the patient will meet with the physician before surgery for an explanatory interview and subsequent signing of informed consent.

INTERVENTIONS:
Other: active informed consent — new preoperative information method, based on multimedia tools and on the objective control of understanding by the patient candidate for vertebral or urological surgery.
  Arms: active informed consent

SUMMARY:
This is an interventional, non-pharmacological, randomized controlled superiority study (RCT), multicenter, open label, parallel group.

The aim is to evaluate the effectiveness of a new preoperative information method, based on multimedia tools and on the objective control of understanding by the patient candidate for spinal or urological surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years (with full legal capacity to consent).
* Scheduled for elective surgery in one of the two domains: spinal surgery or radical prostatectomy in the waiting list of our centers.
* Ability to comprehend Italian language.
* Basic computer or internet access skills. Patients (or their family members) should have the ability to access multimedia content.

Exclusion Criteria:

* Patients under age: minors.
* Inability to provide informed consent or self-determination (significant cognitive impairment, severe mental illness, or decisional incapacity that would prevent them from understanding the consent materials or participating in the decision-making).
* Urgent or emergency surgery cases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | baseline (T0), discharge (T1), 2 months follow-up (T2) and 6 months follow-up (T3)
  The primary outcome of the study will be measured: - by means of the Client Satisfaction Questionnaire, which provides a patient satisfaction score with a range from a minimum of 8 points (completely dissatisfied) to a maximum of 32 points (completely satisfied).

SECONDARY OUTCOMES:
Comprehension Questionnaire | baseline (T0), discharge (T1), 2 months follow-up (T2) and 6 months follow-up (T3)
  procedure-specific assessment tool designed ad-hoc to evaluate a patient's knowledge and understanding of the planned procedure and associated risks/alternatives.
Depression Anxiety Stress Scales (DASS-21) | baseline (T0), discharge (T1), 2 months follow-up (T2) and 6 months follow-up (T3)
  is a 21-item self-report questionnaire designed to assess the severity of depression, anxiety, and stress symptoms over the past week
Numeric Rating Scale (NRS) | baseline (T0), discharge (T1), 2 months follow-up (T2) and 6 months follow-up (T3)
  is a simple self-report measure in which patients rate their current pain intensity on an scale from 0 ("no pain") to 10 ("worst imaginable pain").
Oswestry Disability Index (ODI) | baseline (T0), discharge (T1), 2 months follow-up (T2) and 6 months follow-up (T3)
  self-administered questionnaire that assesses the degree of disability and functional impairment across ten daily-activity domains.
International Prostate Symptom Score (IPSS) | baseline (T0), discharge (T1), 2 months follow-up (T2) and 6 months follow-up (T3)
  Only for Urology patients: 7-item questionnaire that evaluates the severity of lower urinary tract symptoms and their impact on quality of life.
International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) | baseline (T0), discharge (T1), 2 months follow-up (T2) and 6 months follow-up (T3)
  Only for Urology patients: short, patient-completed questionnaire that measures the frequency, severity, and impact of urinary incontinence on quality of life.
International Index of Erectile Function (IIEF-5 ) | baseline (T0), discharge (T1), 2 months follow-up (T2) and 6 months follow-up (T3)
  Only for Urology patients: brief, 5-item self-report measure used to assess erectile function and screen for erectile dysfunction severity
Rate of Patients Declining Spine Surgery (Opt-Out Rate) | baseline (T0)
  The proportion of patients in spine surgery population, who, after receiving full information, choose not to proceed with the planned surgery.
Medico-Legal Outcomes | baseline (T0), discharge (T1), 2 months follow-up (T2) and 6 months follow-up (T3).
  For each group, we will track through hospital records the number of medicolegal complaints or claims filed by patients, specifically those alleging inadequate informed consent or unexpected outcomes, related to their surgery within the follow-up period. The outcome will be reported as the count (or proportion of patients) with such complaints in each arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kinnersley P, Phillips K, Savage K, Kelly MJ, Farrell E, Morgan B, Whistance R, Lewis V, Mann MK, Stephens BL, Blazeby J, Elwyn G, Edwards AG. Interventions to promote informed consent for patients undergoing surgical and other invasive healthcare procedures. Cochrane Database Syst Rev. 2013 Jul 6;2013(7):CD009445. doi: 10.1002/14651858.CD009445.pub2. PMID 23832767
- [Result] Glaser J, Nouri S, Fernandez A, Sudore RL, Schillinger D, Klein-Fedyshin M, Schenker Y. Interventions to Improve Patient Comprehension in Informed Consent for Medical and Surgical Procedures: An Updated Systematic Review. Med Decis Making. 2020 Feb;40(2):119-143. doi: 10.1177/0272989X19896348. Epub 2020 Jan 16. PMID 31948345
- [Result] Nathe JM, Krakow EF. The Challenges of Informed Consent in High-Stakes, Randomized Oncology Trials: A Systematic Review. MDM Policy Pract. 2019 Mar 28;4(1):2381468319840322. doi: 10.1177/2381468319840322. eCollection 2019 Jan-Jun. PMID 30944886
- [Result] Luhnen J, Muhlhauser I, Steckelberg A. The Quality of Informed Consent Forms-a Systematic Review and Critical Analysis. Dtsch Arztebl Int. 2018 Jun 1;115(22):377-383. doi: 10.3238/arztebl.2018.0377. PMID 29932049